CLINICAL TRIAL: NCT06597929
Title: The Effectiveness of Moderate-vigorous Intermittent Lifestyle Physical Activity and Health Education to Increase Intense Physical Activity in Stroke Survivors: a Pragmatic Randomised Controlled Trial (MV-ILPA-stroke)
Brief Title: Moderate-vigorous Intermittent Physical Activity (M-VILPA) in Stroke
Acronym: PA-stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, PhD, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-VILPA-stroke
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Physical Inactivity; Stroke
Keywords: Physical activity; Stroke; Moderate-vigorous physical activity
MeSH Terms: conditions — Sedentary Behavior; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus the MV-ILPA and education program. (Experimental): The experimental group will receive usual care plus the MV-ILPA and education program. First, a physiotherapist will conduct a face-to-face session with the patients detailing the health benefits of moderate to vigorous PA and the negative effects of not including it in their daily lives. Patients will receive a booklet with all the key information. Secondly, participants will take the MV-ILPA program.
  Interventions: Other: Moderate-vigorous physical activity
- Usual care (Active Comparator): Usual care: appointments with the treating neurologist, medication, conventional physiotherapy (two/three times a week, including stretching, strength, and balance training), occupational therapy, and speech therapy if required.
  Interventions: Other: Moderate-vigorous physical activity

INTERVENTIONS:
Other: Moderate-vigorous physical activity — The experimental group will receive usual care plus the MV-ILPA and education program. First, a physiotherapist will conduct a face-to-face session with the patients detailing the health benefits of moderate to vigorous PA and the negative effects of not including it in their daily lives. Patients will receive a booklet with all the key information. Secondly, participants will take the MV-ILPA program. This program consists of completing 4 length-standardised moderate-to-vigorous intense bouts per day (3 minutes each) of activities of daily living (sit-to-stand, going up/down stairs, walking fast indoors, and walking up small slopes) every day for 12 weeks. Once per week for 12 weeks, a physiotherapist will go to the patient's home for a face-to-face session or videoconference. This physiotherapist will foster participants' independence and self-management. The PA intensity will be increased weekly by increasing the execution speed and including weights.
  Other Names: Moderate-vigorous exercise

SUMMARY:
Stroke is the leading cause of disability in Spain. Additionally, it is the second leading cause of death in women and the third in both sexes. Regular physical activity (PA) helps prevent and manage stroke. It also helps with hypertension, maintains a healthy body weight, and improves mental health, quality of life, and well-being. PA plays a prominent role in inpatient care after stroke. However, stroke survivors become more sedentary when discharged from the hospital. They have muscle weakness, reduced balance, and fatigue. Consequently, PA levels of community-dwelling post-stroke individuals remain lower than their age-matched counterparts. Continued PA can help this population maintain and improve physical function, and reduce long-term functional limitations, and mortality risk.

DETAILED DESCRIPTION:
Previous studies that performed a comparative analysis of physical activity between individuals with and without stroke have consistently reported that stroke survivors tend to spend less time in moderate to vigorous physical activity The 2021 AHA guideline recommends smaller sessions of PA, with suggestions such as 10 minutes of moderate activity, 4 times a week, or 20 minutes of vigorous activity twice a week. This contrasts the weekly physical activity recommendations in 2011 (30 minutes of moderate to vigorous, 1 to 3 times) and 2014 (40 minutes of moderate to vigorous, 3 to 4 times). We hypothesise that older stroke survivors are physically active more frequently but for smaller durations than younger stroke survivors who are physically active for longer durations but less regularly. Understanding these subtle changes will not only help to tailor physical activity interventions based on specific recommendations but also help design future recommendations.

Moderate-to-vigorous PA could be an adequate approach for stroke survivors as it requires less time to achieve the same benefits as light PA. More concretely, a new concept called moderate-to-vigorous intermittent lifestyle physical activity (MV-ILPA) has recently emerged for adults who do not habitually exercise in their leisure time. MV-ILPA refers to brief and sporadic bouts of moderate-vigorous intensity PA performed as part of the activities of daily living, such as bursts of very fast walking, sitting and standing up from a chair, or stair climbing. MV-ILPA is associated with a substantially lower risk of all-cause cardiovascular disease and cancer mortality. However, there is no evidence to directly support the potential benefits of MV-ILPA in the elderly post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥57 in the late subacute phase post-stroke.
* who live in the community
* whose clinician confirmed a diagnosis of stroke (ischaemic/haemorrhagic)
* discharged from hospital inpatient regimen
* with independent mobility skills (Barthel Index ≥ 40 points).

Exclusion Criteria:

• other neurological diseases (e.g. Parkinson disease) or severe lower limb injuries.

Min Age: 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The amount of moderate-vigorous intense physical activity (PA). | The measurements will be performed during the week before Day 0 and Month 3.
  All participants will be monitored with a 3-axial accelerometer (strapped on the thigh) for 7 days to record their total daily movement counts and the minutes of moderate-to-vigorous-intensity PA.

SECONDARY OUTCOMES:
Lower limb peak power | Day 0 and Month 3
  The participants were instructed to rise from the chair, without armrests, as fast and powerful as possible, reaching a fully standing erect position without lifting their feet and sit back down as quickly as possible. Three attempts were given interspersed by 30-60 s. The attempt with the highest peak power was selected for further analyses. It is measured in Watts.Higher peak power means better outcome.
Balance | Day 0 and Month 3
  It will be assess by Berg Balance Scale, 0-56 points higher scores means better outcome
Gait speed | Day 0 and Month 3
  4-metre walk test, less time mean better outcome
Fatigue | Day 0 and Month 3
  Fatigue Severity Scale, a 9-item questionnaire The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher score means worse outcome.
Quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. | Day 0 and Month 3
  It will be assess by EuroQol 5-dimension 5-level. Each dimension is described by 5 possible levels, scoring from 0 to 25 points. Higher score means worse outcome.
Degree of disability | Day 0 and Month 3
  Modified-Rankin Scale, single-item global outcomes rating scale, from 0 to 5. Higher score means worse outcome.
Stroke recurrence | Day 0 and Month 3
  yes/no, date
Death | Day 0 and Month 3
  yes/no, date
Falls | Day 0 and Month 3
  yes/no, date

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Cabanas-Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabanas-Valdes R, Garcia-Rueda L, Salgueiro C, Perez-Bellmunt A, Rodriguez-Sanz J, Lopez-de-Celis C. Assessment of the 4-meter walk test test-retest reliability and concurrent validity and its correlation with the five sit-to-stand test in chronic ambulatory stroke survivors. Gait Posture. 2023 Mar;101:8-13. doi: 10.1016/j.gaitpost.2023.01.014. Epub 2023 Jan 20. PMID 36696822
- [Background] Kwakkel G, Stinear C, Essers B, Munoz-Novoa M, Branscheidt M, Cabanas-Valdes R, Lakicevic S, Lampropoulou S, Luft AR, Marque P, Moore SA, Solomon JM, Swinnen E, Turolla A, Alt Murphy M, Verheyden G. Motor rehabilitation after stroke: European Stroke Organisation (ESO) consensus-based definition and guiding framework. Eur Stroke J. 2023 Dec;8(4):880-894. doi: 10.1177/23969873231191304. Epub 2023 Aug 7. PMID 37548025
- [Background] Goncalves S, Le Bourvellec M, Duclos NC, Mandigout S. Recommended moderate to vigorous physical activity levels for people in the chronic phase of stroke can be achieved in outpatient physiotherapy: a multicentre observational study. Top Stroke Rehabil. 2025 Apr;32(3):219-228. doi: 10.1080/10749357.2024.2392447. Epub 2024 Aug 22. PMID 39172127
- [Background] Boyne P, Billinger SA, Reisman DS, Awosika OO, Buckley S, Burson J, Carl D, DeLange M, Doren S, Earnest M, Gerson M, Henry M, Horning A, Khoury JC, Kissela BM, Laughlin A, McCartney K, McQuaid T, Miller A, Moores A, Palmer JA, Sucharew H, Thompson ED, Wagner E, Ward J, Wasik EP, Whitaker AA, Wright H, Dunning K. Optimal Intensity and Duration of Walking Rehabilitation in Patients With Chronic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Apr 1;80(4):342-351. doi: 10.1001/jamaneurol.2023.0033. PMID 36822187
- [Background] Stamatakis E, Ahmadi MN, Friedenreich CM, Blodgett JM, Koster A, Holtermann A, Atkin A, Rangul V, Sherar LB, Teixeira-Pinto A, Ekelund U, Lee IM, Hamer M. Vigorous Intermittent Lifestyle Physical Activity and Cancer Incidence Among Nonexercising Adults: The UK Biobank Accelerometry Study. JAMA Oncol. 2023 Sep 1;9(9):1255-1259. doi: 10.1001/jamaoncol.2023.1830. PMID 37498576